CLINICAL TRIAL: NCT00679328
Title: Study #91-01 - A Randomized Study of the Stryker OP Device vs. Bone Autograft for the Treatment of Tibial Nonunions
Brief Title: OP Device vs. Bone Autograft for the Treatment of Tibial Nonunions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Biotech Corporation (Industry)
Responsible Party: Shinichi Torii, Olympus Biotech
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91-01; TR-0056
Record Dates: First submitted 2008-05-13; First posted 2008-05-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Tibial Nonunions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Surgical implantation of OP-1
  Interventions: Device: Surgical implantation of OP-1 device or autograft bone graft material
- 2 (Active Comparator): Surgical implantation of bone graft material
  Interventions: Device: Surgical implantation of OP-1 device or autograft bone graft material

INTERVENTIONS:
Device: Surgical implantation of OP-1 device or autograft bone graft material — Surgical implantation of OP-1 device or autograft bone graft material

SUMMARY:
This study is to evaluate the safety and effectiveness of the OP device for the treatment of nonunion bone fractures and to compare the healing rates of the OP Device to that of autograft.

DETAILED DESCRIPTION:
This study is to evaluate the safety and effectiveness of the OP device for the treatment of nonunion bone fractures and to compare the clinical safety and effectiveness (healing rates) of the OP Device to that of traditional bone autografts to repair nonunions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must show radiographic skeletal maturity
2. Documented evidence of previous fracture management
3. Nonunion in the tibia and candidate to receive bone autografts and intramedullary (IM) Nail fixation
4. Nonunion gap must not exceed half the diameter of the bone at the site of fracture, as assessed radiographically prior to study treatment

Exclusion Criteria:

1. Patients who do not have adequate vascularity to permit healing
2. Patients with inadequate skin coverage
3. Patients with chronic use of steroidal medications
4. Patients with active infection systemically or at the site of nonunion.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 1992-02; Primary Completion 1996-08 (Actual); Study Completion 1999-12 (Actual)

PRIMARY OUTCOMES:
No further retreatment of the surgical site, function and pain at the site of the nonunion, evidence of bridging. | 3, 6, 9, 12, 24 months

SECONDARY OUTCOMES:
Medical events, treatment related events, laboratory tests, medication use. | 3, 6, 9, 12, 24 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Mesa, Arizona
  - Modesto, California
  - San Diego, California
  - Stanford, California
  - Denver, Colorado
  - Fort Carson, Colorado
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - New Orleans, Louisiana
  - Detroit, Michigan
  - St Louis, Missouri
  - New York, New York
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Galveston, Texas
  - Lubbock, Texas